CLINICAL TRIAL: NCT05292729
Title: Cognitive Function and Brain Connectivity in Carotid Artery Stenting Patients:a Rs-fMRI Study
Brief Title: Cognitive Function and Brain Connectivity in CAS Patients:a Rs-fMRI Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 3.0T rs-fMRI
Record Dates: First submitted 2021-12-27; First posted 2022-03-23 (Actual); Last update posted 2022-03-23 (Actual); Status verified 2021-12

CONDITIONS: MRI, Functional; Carotid Artery Stenosis
Keywords: resting state; MRI; carotid artery stenting; cognition
MeSH Terms: conditions — Carotid Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This is a prospective study aimed to explore the changes of cognitive function after surgery for CAS and the correlation with brain connectivity, in order to look for the clinical biomarkers to predict the carotid stent implantation for patients which can effect the cognition

DETAILED DESCRIPTION:
Carotid artery stenting (CAS) can significantly decrease the incidence of ischemic stroke in patients with severe carotid artery stenosis has been confirmed in large randomized controlled studies (1, 2).Previous studies showed carotid artery stenosis is closely related to cognitive dysfunction, including asymptomatic carotid artery stenosis(≥70%).Cognitive impairment is one of the most serious problem facing the elderly. The impact on cognitive function in patients with CAS has been discussed by many researchers, however the effect still remained conflicting.

In past few years, several imaging techniques, such as resting-state functional MRI (R-fMRI), had been increasingly used to study cognitive impairment in humans. In this study, we evaluated the cognition performance in severe carotid artery stenosis patients undergoing CAS and explored the mechanisms underlying the cognition changes by the Rs-fMRI.

Inclusion criteria:

* age between 55 years and 80 years
* unilateral internal carotid artery stenotic degree ≥ 70%
* right-hand-dominant
* free of dementia, and depression
* modified Rankin Scale: 0 or 1
* education ≥6 years
* obtained written informed consent.

Exclusion criteria:

* contralateral internal carotid artery stenosis ≥ 50%
* posterior circulation diseases
* MMSE < 26, which is a cut-off value for mild cognitive impairment
* severe systemic diseases and neuropsychiatric diseases (such as congestive heart failure)
* any contraindications for MRI scan (e.g., metal implants)
* Non atherosclerotic stenosis, such as dissection, vasculitis.

ELIGIBILITY:
Inclusion Criteria:

* age between 55 years and 80 years
* unilateral internal carotid artery stenotic degree ≥ 70%
* right-hand-dominant
* free of stroke, TIA, dementia, and depression
* modified Rankin Scale: 0 or 1
* education ≥6 years
* obtained written informed consent.

Exclusion Criteria:

* contralateral internal carotid artery stenosis ≥ 50%
* posterior circulation diseases
* MMSE < 26, which is a cut-off value for mild cognitive impairment
* severe systemic diseases and neuropsychiatric diseases (such as congestive heart failure and history of stroke)
* any contraindications for MRI scan (e.g., metal implants)

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: consecutive enrolled patients with carotid artery stenosis who undergoing carotid artery stenting
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
Montreal Cognitive Assessment, MOCA | before CAS(within 1 week)
  use MOCA to assess the cognition before CAS
Mini-mental State Examination，MMSE | before CAS(within 1 week)
  use MMSE to assess the cognition before CAS
Montreal Cognitive Assessment, MOCA | 3 months after CAS
  use MOCA to assess the cognition after CAS
Mini-mental State Examination，MMSE | 3 months after CAS
  use MMSE to assess the cognition after CAS

SECONDARY OUTCOMES:
Digit Symbol Test | before CAS(within 1 week)
  use to assess the cognition before CAS
Digit Symbol Test | 3 months after CAS
  use to assess the cognition after CAS
Trail Making Test A/B | before CAS(within 1 week)
  use to assess the cognition before CAS
Trail Making Test A/B | 3 months after CAS
  use to assess the cognition after CAS
digital span test | before CAS(within 1 week)
  use to assess the cognition before CAS
digital span test | 3 months after CAS
  use to assess the cognition after CAS

CONTACTS AND LOCATIONS:
Overall Officials: Benyan Luo, PhD, Principal Investigator — Zhejiang University
Locations (1):
- the first affiliated hospital of Zhejiang university, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ji R, Zhang S, Chen H, Deng C, Xu Z, Zhang J, Luo B. Impact of Endovascular Revascularization on Functional Connectivity and Cognition in Symptomatic Chronic Internal Carotid Artery Occlusion Patients: A Preliminary Exploratory Study. J Integr Neurosci. 2025 Apr 24;24(4):36330. doi: 10.31083/JIN36330. PMID 40302264